CLINICAL TRIAL: NCT04984616
Title: Effect of Statins (Atorvastatin) on Inflammation and Cardiac Function in Patients with Chronic Chagas Disease: Pathophysiological Studies in a Multicenter Proof-of-concept
Brief Title: Atorvastatin on Inflammation and Cardiac Function in Chronic Chagas Disease
Acronym: ATOCHA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The recruitment rate in all centers was extremely low. The number of participants failed to reach a statistically significant minimum.
Sponsor: Juan D. Maya (Other)
Responsible Party: Sponsor-Investigator, Juan D. Maya, Full Professor, University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1267-3513
Record Dates: First submitted 2021-06-29; First posted 2021-07-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Chronic Chagas Disease
Keywords: Chagas Disease; Atorvastatin; Inflammation
MeSH Terms: conditions — Chagas Disease; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ATORVASTATIN 40 (Experimental): 40 mg Atorvastatin/day for 120 days P.O.
  Interventions: Drug: 40 mg Atorvastatin/day for 120 days P.O.
- ATORVASTATIN 80 (Experimental): 80 mg Atorvastatin/day for 120 days P.O.
  Interventions: Drug: Atorvastatin 80
- Placebo (Placebo Comparator): Placebo/day for 120 days P.O.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 40 mg Atorvastatin/day for 120 days P.O. — Oral administration of Atorvastatin 40 mg/daily for 120 days
  Arms: ATORVASTATIN 40
Drug: Atorvastatin 80 — Oral administration of Atorvastatin 80 mg/daily for 120 days
  Arms: ATORVASTATIN 80
Drug: Placebo — Oral administration of Placebo daily for 120 days
  Arms: Placebo

SUMMARY:
Chagas Disease, caused by the parasite Trypanosoma cruzi afflicts 7 million people in Latin America, and due to migration, abroad. The diagnosis lies in clinical suspicion and serologic detection of antibodies. Cardiac evaluation is essential because complications, including heart failure and arrhythmias, are the main causes of disability and death. Heart involvement is explained by a parasite-dependent, immune-mediated myocardial and microvascular injuries.

Current treatment includes the administration of nifurtimox or benznidazole, although in the chronic phase their efficacy is low and may induce severe adverse events, forcing the suspension of the therapy. Therefore, finding innovative approaches to improve the efficacy of the current antichagasic drugs by modifying the inflammatory response would render the current treatment more effective.

Pre-clinical evidence supports the idea that the cholesterol-lowering statin drugs, such as atorvastatin, may contribute to decrease cardiac inflammation, reduce endothelial activation, and improve cardiac function. Atorvastatin therapeutic and safety profiles are well known, as is its mechanism of action, shared by the other members of the statin class.

This trial aims at evaluating whether atorvastatin, in combination with antichagasic therapy, is safe and more efficacious in reducing general inflammation than an antiparasitic therapy alone, by improving endothelial and cardiac functions.

This proof-of-concept trial will be double-blinded, randomized, and multicentered with a phase II design. To achieve this aim, it will be evaluated the efficacy of the combination of atorvastatin and antichagasic therapy (nifurtimox or benznidazole) to reduce inflammatory cytokine plasma levels, soluble endothelial cell adhesion molecules, and confirm the improvement of the cardiac function by electrocardiogram and two-dimensional echocardiogram.

The trial will set the safety and tolerability of the combination of atorvastatin with antichagasic therapy by monitoring the incidence of adverse events and discontinuation of the therapy.

This trial will be conducted with a sample size of 300 adult patients in four hospitals located in Santiago and Valparaiso, Chile.

DETAILED DESCRIPTION:
Chagas disease (CD) afflicts 7 million people in 21 endemic countries in Latin America and is increasing in non-endemic countries due to migration. Control programs are discontinuous and current therapy is limited due to low efficacy.

Different biomarkers have been proposed to evaluate progression, prognosis, or response to treatment; but, none has demonstrated sufficient specificity to be a gold standard for CD diagnosis. However, brain natriuretic peptide (BNP) and cardiac troponin T (cTnT) have been proposed as useful biomarkers to predict progress towards left ventricular dysfunction.

Chronic Chagas Cardiomyopathy (CCC) is caused by a parasite-dependent, immune-mediated myocardial damage, which is the most critical determinant of the disease where the T helper 1/T helper 2 /T regulatory response is a crucial feature, where the equilibrium between excessive pro-inflammatory (Interferon-γ, tumor necrosis factor-α, IL-1β) and anti-inflammatory (IL-4, IL-10) cytokines is critical for cardiac damage development. Also, microvascular abnormalities and ischemia secondary to platelet activation and endothelial dysfunction, as evidenced by increases in cell adhesion molecules Intercellular Adhesion Molecule type 1 (ICAM-1), Vascular Cell Adhesion Molecule (VCAM), and E-selectin, including their soluble forms.

Treatment of CCC and improvement strategies: In Chile, the etiologic treatment of CD in Chile is done with 5-10 mg/kg/day nifurtimox (NFX) or 5 mg/kg/day benznidazole (BZD) for 60 days. Drug therapy during the acute phase, congenital disease, and early indeterminate phase has a satisfactory efficacy and is considered curative. However, it is more difficult to declare a cure for chronic infection because current evidence of drug efficacy in this phase is weak or controversial, especially when mortality is considered.

There are molecules involved in the natural resolution of inflammation. These specialized pro-resolving mediators include several lipids that control the magnitude and duration of local inflammation. These lipids are derived from essential fatty acids present in the plasma membrane, such as arachidonic acid or docosahexaenoic acid. Interestingly, aspirin and cholesterol-lowering statins, including atorvastatin can induce the synthesis of such molecules.

Thus, a combination of trypanocidal drugs and those inducing resolution of the inflammatory process derived from parasite persistence could be a sound therapeutic strategy to prevent chronic consequences of CD.

There is a general agreement that adults with chronic indeterminate CD are the population with the most urgent requirements for the development of new treatments because of the highest disease burden to these patients. Thus, improving the host's factors (e.g., the immune reaction elicited) may increase the efficacy of the conventional antichagasic therapy, probably by a decrease in the dose, a decrease in its duration, or both. The therapeutic and safety profiles of atorvastatin are well known, as is its mechanism of action and pharmacological actions, including the anti-inflammatory properties, shared by the other members of the statin class. Importantly, due to the low incidence of severe adverse events and efficacy, is one of the most widely used statins today. 20-80 mg/day atorvastatin is used to decrease the so-called LDL cholesterol involved in the pathogenesis of atherosclerotic cardiovascular disease.

Thus, this trial aims at evaluating whether atorvastatin, in combination with antichagasic therapy, is safe and more efficacious in reducing general inflammation than an antiparasitic therapy alone, by improving endothelial and cardiac functions.

This proof-of-concept trial will be double-blinded, randomized, and multicentered with a phase II design. To achieve this aim, it will be evaluated the efficacy of the combination of atorvastatin and antichagasic therapy (nifurtimox or benznidazole) to reduce inflammatory cytokine plasma levels, soluble endothelial cell adhesion molecules, and confirm the improvement of the cardiac function by electrocardiogram and two-dimensional echocardiogram.

This clinical trial will be conducted in four centers located in the cities of Santiago and Valparaiso, Chile. In all those centers, well-established Programs for Chagas Control (PCC) are ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 18 and younger than 50 years,
* with a weight higher than 40 kg
* Positive conventional confirmatory serology for T. cruzi infection from the NAtional Public Health institute (ISPCH), and
* A positive qPCR
* Have normal laboratory test values for the following parameters: total white blood cell count, platelet count, creatine kinase (CK), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin or creatinine, or a gamma-glutamyl transferase (GGT) > 2 times the upper limit of normal (X ULN);
* Women of reproductive age must have a negative serum pregnancy test, must not be breastfeeding, and must consistently use a highly effective contraceptive method throughout the treatment phase
* Ability to comply with all protocol-specified follow-up tests and visits and have a permanent address;
* Signed written informed consent form

Exclusion Criteria:

* Signs and symptoms of the digestive form of Chagas Disease;
* Chronic cardiac Chagas Disease stage II or higher;
* Acute or chronic health conditions such as acute infections, history of HIV infection, diabetes, liver and kidney disease;
* Hypothyroidism
* Family history of muscle disorders
* Pre-existing heart disease unrelated to Chagas disease;
* Formal contraindication to receive nifurtimox or benznidazole,
* Known history of hypersensitivity, allergy or severe adverse reactions to atorvastatin, benznidazole or nifurtimox;
* History of previous treatment for Chagas Disease;
* History of prior treatment with atorvastatin, lovastatin, rosuvastatin, simvastatin or any other statin;
* Any concomitant use of antimicrobial agents;
* History of alcohol or drug abuse;
* Any condition that precludes oral medication;
* Concomitant or intended use of CYP3A4 modifiers;
* Medical history of familial short QT syndrome or concomitant therapy with medications that may shorten the QT interval.
* Abnormal laboratory test values for the following parameters: total white blood cell count, platelet count, creatine kinase (CK), alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin or creatinine, or a gamma-glutamyl transferase (GGT) > 2 times the upper limit of normal (X ULN);
* Being pregnant or breastfeeding
* Refusing to use a highly effective contraceptive method during the treatment phase.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients that present a change in the phase of the chronic cardiomyopathy | Twelve months
  To evaluate whether the effect of atorvastatin in combination with antiparasitic therapy (NFX or BZD), more effective than antiparasitic therapy alone in preventing the onset of cardiac disorders as determined by non-progression in the phase from the A-phase according to the I Latin American Guidelines for the diagnosis and treatment of Chagas cardiomyopathy (Andrade et al, Arq Bras Cardiol 2011;97 Suppl 3:1-48.).

SECONDARY OUTCOMES:
plasma levels of cytokines (pg/mL) | Twelve months
  Plasma levels of the tumor necrosis factor -α, interferon -γ, IL-10, IL-1B, IL-4, and IL-17A cytokines will be determined by a multiplex analysis
Plasma levels of endothelial adhesion molecules (pg/mL) | Twelve months
  Plasma levels of the soluble forms of Intercellular Cell Adhesion Molecule-1, Vascular Cell Adhesion Molecule-1, and E-selectin, as determined by a multiplex analysis
Proportion of patients with change in heart rate measured by electrocardiographic examination | Twelve months
  Percentage of patients in the treatment arms that present changes in cardiac rate as compared with the placebo arm
Proportion of patients with changes in the QT interval duration (milliseconds) | Twelve months
  Percentage of patients in the treatment arms that present changes in repolarization, as determined by the QT interval duration in the electrocardiogram, when compared with the placebo arm
Proportion of patients with abnormalities in ventricular electrical conduction determined by the duration of the QRS interval (milliseconds) | Twelve months
  Percentage of patients in the treatment arms that present changes in ventricular conduction, as determined by QRS interval duration in the electrocardiogram, when compared with the placebo arm
Proportion of patients with alterations in ventricular function as measured by changes in the ejection fraction percentage estimated by echocardiography | Twelve months
  Percentage of patients in the treatment arms that present changes in ventricular function, as determined by ejection fraction calculated using echocardiography analysis, when compared with the placebo arm.
Plasma levels of Cardiac function biomarkers (pg/mL) | Twelve months
  Cardiac functional damage evidenced by a change in the plasma levels of brain natriuretic peptide (BNP) and cardiac troponin T (cTnT)
Parasite load in a blood sample (number of parasites/mL) | Twelve months
  To determine the parasitic load in blood by quantitative polymerase chain reaction assay (qPCR)
Incidence of severe adverse events | Twelve months
  To evaluate the incidence of treatment discontinuation due to severe Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Juan D. Maya, Ph.D., Principal Investigator — Full Professor
Locations (4):
- Chile (4):
  - Hospital San Martin, Quillota, Región de Valparaíso
  - Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso
  - Hospital Felix Bulnes, Quinta Normal, Santiago Metropolitan
  - Hospital San Juan de Dios, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: Undecided
The study protocol and the Clinical Study Report will be available as supporting information alongside all publications derived from this study.
  By incorporating the Individual Participant Data on a repository after an embargo period of one year after the last patient is recruited

REFERENCES:
- [Derived] Campos-Estrada C, Urarte E, Denegri M, Villalon L, Gonzalez-Herrera F, Kemmerling U, Maya JD. Effect of statins on inflammation and cardiac function in patients with chronic Chagas disease: A protocol for pathophysiological studies in a multicenter, placebo-controlled, proof-of-concept phase II trial. PLoS One. 2023 Jan 13;18(1):e0280335. doi: 10.1371/journal.pone.0280335. eCollection 2023. PMID 36638112